CLINICAL TRIAL: NCT06175624
Title: Effect of Non-Surgical Periodontal Treatment on Gingival Crevicular Fluid and Serum Biomarker Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burcu KARADUMAN, Proffesor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-KAEK-79-23-07
Record Dates: First submitted 2023-12-04; First posted 2023-12-19 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis; Gingivitis; Healthy
Keywords: Periodontitis; Periodontal Therapy; Biomarker
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Intervention Model Description: 25 patients with periodontitis, 25 with gingivitis and 25 healthy periodontals (total of 75 individuals) will be included in our study. At the beginning of the study, periodontal clinical measurements (gingival index, plaque index, probing depth, gingival recession, clinical attachment level, and bleeding on probing), serum and gingival crevicular fluid samples will be taken from all individuals. Non-surgical periodontal treatment will be applied in quadrant wise within 2 weeks to individuals with gingivitis and periodontitis. 12 weeks after treatment; the clinical measurements and the collection of serum and gingival crevicular fluid will be repeated. Biomarkers in serum and gingival crevicular fluid samples will be examined by ELISA.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinical Healthy (Active Comparator): Our study will include 25 people with clinically healthy patients.
  Interventions: Other: Clinically Helathy
- Gingivitis (Experimental): Our study will include 25 people with gingivitis patients.
  Interventions: Other: Gingivitis
- Periodontitis (Experimental): Our study will include 25 people with periodontitis patients.
  Interventions: Other: Periodontitis

INTERVENTIONS:
Other: Clinically Helathy — Our study will include 25 people with clinically healthy patients.
  Gingival crevicular fluid and serum will be collected during the clinical measurements Biomarkers in serum and gingival crevicular fluid samples will be examined by ELISA.
  CTRP-1 levels will be examined to evaluate the effects of periodontal treatment in periodontal health, gingivitis and periodontitis.
  Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and sample will be taken from all individuals at the beginning of the study.
  Arms: Clinical Healthy
Other: Gingivitis — Our study will include 25 people with gingivitis patients.
  Gingival crevicular fluid and serum will be collected during the clinical measurements Biomarkers in serum and gingival crevicular fluid samples will be examined by ELISA.
  CTRP-1 levels will be examined to evaluate the effects of periodontal treatment in periodontal health, gingivitis and periodontitis.
  Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and sample will be taken from all individuals at the beginning of the study.
  Arms: Gingivitis
Other: Periodontitis — Our study will include 25 people with periodontitis patients.
  Non-surgical periodontal treatment will be applied to individuals with periodontitis, serum and gingival crevicular fluid samples will be collected before the treatment, clinical measurements and gingival crevicular fluid and serum collection will be repeated 12 weeks after the treatment. CTRP-1 analysis will be performed by ELISA.
  CTRP-1 levels will be examined to evaluate the effects of periodontal treatment in periodontal health, gingivitis and periodontitis.
  Clinical measurements (Plaque index, probing depth, gingival recession, clinical attachment level, bleeding on probing) and salivary sample will be taken from all individuals at the beginning of the study.
  Arms: Periodontitis

SUMMARY:
Periodontal diseases are one of the most common inflammatory diseases. Periodontitis results from products and antigens of microorganisms, which stimulates the innate immune system and local inflammatory response; characterized by gingival inflammation, attachment loss, and alveolar bone destruction. Molecules that play a role in the pathogenesis of periodontal disease can be used as biomarkers in the early diagnosis of periodontitis, in determining the rate of periodontal destruction, and in evaluating the response to periodontal treatment.

CTRPs (C1q/TNF-related proteins), which are adiponectin paralogs, are involved in inflammation, lipid, and glucose metabolism, as well as physiological and pathological processes like vasodilation. CTRP-1 is a glycoprotein belonging to the CTRP family that can be detected in serum in the presence of certain antibodies. Serum CTRP-1 levels increase in type 2 diabetes, prediabetes, coronary artery diseases, congestive heart failure, and atherosclerosis. Lipopolysaccharides found in Gram-negative bacteria cell walls stimulate the production of inflammatory cytokines such as tumor necrosis factor (TNF)-α and interleukin (IL)-1 β, as well as indirectly increasing the production of CTRP-1. CTRP-1 is a therapeutic target in many inflammatory diseases, including periodontal diseases. However, there are no clinical studies on the role of CTRP-1 in the pathogenesis of periodontal disease. Based on these findings, the goal of our research is to examine the effects of periodontal disease on CTRP-1, IL-10, and TNF-α levels in serum and gingival crevicular fluid samples taken before and after periodontal treatment from periodontally healthy individuals and individuals with gingivitis and periodontitis, and also determine whether CTRP-1 is a potential biomarker that can be used in the diagnosis of periodontal disease.

25 patients with periodontitis, 25 with gingivitis and 25 healthy periodontals (total of 75 individuals) will be included in our study. At the beginning of the study, periodontal clinical measurements (gingival index, plaque index, probing depth, gingival recession, clinical attachment level, and bleeding on probing), serum and gingival crevicular fluid samples will be taken from all individuals. Non-surgical periodontal treatment will be applied in quadrant wise within 2 weeks to individuals with gingivitis and periodontitis. 12 weeks after treatment; the clinical measurements and the collection of serum and gingival crevicular fluid will be repeated. Biomarkers in serum and gingival crevicular fluid samples will be examined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal healthy group
* Stage III Grade B Periodontitis Group
* To meet the above-mentioned periodontal health and disease criteria

Exclusion Criteria:

* Periodontal tissues, periodontal disease course, periodontal application training and to have,
* Chronic alcohol and cigarette use,
* Oral contraceptive use, pregnancy, pregnant,
* Use of antibiotics or anti-inflammatory drugs within the last 6 months,
* Having undergone periodontal treatment in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Examination of CTRP-1 levels of periodontal disease and clinically healthy | up to 1 year
  Examination of CTRP-1 levels, which are stated to be associated with periodontal disease, in gingival crevicular fluid and serum samples obtained from individuals with periodontitis.
Evaluation of the effect of non-surgical periodontal treatment on changes in CTRP-1 level. | up to 1 year
  Evaluation of the effect of non-surgical periodontal treatment on changes in CTRP-1 level.
Comparison biomarkers of study groups. | up to 1 year
  Comparison of gingival crevicular fluid and serum samples taken before treatment in individuals with periodontitis in terms of CTRP-1 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversity, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided